CLINICAL TRIAL: NCT06319261
Title: Efficacy of Guided Biofilm Therapy (GBT) for Treatment of Deep Periodontal Pockets: A Randomized Clinical Trial
Brief Title: Efficacy of Guided Biofilm Therapy (GBT) for Treatment of Deep Periodontal Pockets.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Reem Hussain Faisal, dentist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 858623
Record Dates: First submitted 2024-03-04; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- guided biofilm therapy group (Active Comparator): Sites treated with guided biofilm therapy.
  Interventions: Procedure: guided biofilm therapy
- conventional root debridement group (Other): Sites treated with conventional manual instrumentation only.
  Interventions: Procedure: root surface debridement

INTERVENTIONS:
Procedure: guided biofilm therapy — Removing plaque and calculus by initially detecting it with a disclosing agent followed by the use of air abrasive powder for the removal of supra and subgingival plaque.
  Arms: guided biofilm therapy group
Procedure: root surface debridement — Removing plaque and calculus by conventional root surface debridement
  Arms: conventional root debridement group

SUMMARY:
the aim of the study is to evaluate the efficacy of guided biofilm therapy (GBT) for treatment of deep periodontal pockets.

the objectives are

1- To compare the change in the clinical periodontal parameters and microbiological parameters by using real time PCR for P. gingivalis, Aggregatibacter actinomycetemcomitans and Filifactor alocis among sites treated by GBT and conventional hand instrumentation after a period of 3 months and to assess the level of the selected periodontal pathogens in deep periodontal pockets and to estimate and compare deep periodontal pockets which need surgery after 3 months of non-surgical treatment by GBT and conventional hand instrumentation.

the hypothesis is whether there are no differences in in the clinical and microbiological parameters among sites treated by GBT and conventional hand instrumentation after a period of 3 months or there are differences in in the clinical and microbiological parameters among sites treated by GBT and conventional hand instrumentation after a period of 3 months.

The participants will be selected on a consecutive basis from patients referred to the Department of Periodontics, College of Dentistry, University of Baghdad.

For each patient, each site will be randomly assigned to either treatment protocol:

1. Sites treated with GBT.
2. Sites treated with conventional manual instrumentation only.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, aged more than 18 years.
2. No history of any systemic diseases.
3. Diagnosed with Stages 3 and 4 periodontitis according to the 2017 World Workshop on the Classification of Periodontal disease.
4. The presence of deep periodontal pocket ≥ 6 mm in two non-adjacent teeth.

Exclusion Criteria:

1. Smokers.
2. Pregnant and lactating mothers.
3. History of any previous subgingival instrumentation in the last 3 months.
4. The use of antibiotics/non-steroidal anti-inflammatory drugs in the last 3 months.
5. Regular use of medication to control systemic illness.
6. The presence of perio-endo lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Periodontal pocket depth (PPD) | 3 months
  PPD will be measured from the gingival margin to the base of the pocket by using the University of North Carolina 15 probe (UNC15) probe to measure the reduction of the pocket depth in millimeters.

SECONDARY OUTCOMES:
Plaque index | 3 months
  Biofilm will be determined using a dichotomous scoring system as present (1) or absent (0) after using a disclosing agent to assess the agreement on the scoring of the biofilm.
Bleeding on probing | 3 months
  Bleeding on probing will be recorded as present (1) or absent (0) after probing all the sites by using UNC15 probe.
Relative attachment level | 3 months
  Relative attachment level will be recorded by making a customized acrylic stent and then measuring the relative attachment level from a fixed point on the stent to the base of the pocket by using UNC15 probe in millimeters.
Changes in the bacterial load | 3 months
  Real time polymerase chain reaction (qPCR) will be used to assess the detection and the quantity of these periodontal pathogens (P.gingivalis, Aggregatibacter actinomycetemcomitans and filifacter alocis) in the subgingival biofilm sample according to the manufacturer's instructions. identification of target bacteria through PCR will be executed using species specific primers.

IPD SHARING:
Plan to Share IPD: Undecided